CLINICAL TRIAL: NCT00612300
Title: The Lokomat Gait Orthosis Compared to Categorized Gait Training by Physical Therapists in Patients Early Post Stroke
Brief Title: Gait Training for Persons With Stroke
Acronym: GTS
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: John Brincks, PT, PhD student, Hammel Neurorehabilitation and Research Center
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 2
Record Dates: First submitted 2008-01-28; First posted 2008-02-11 (Estimated); Last update posted 2010-02-17 (Estimated); Status verified 2010-02

CONDITIONS: Stroke; Middle Cerebral Artery Infarction
Keywords: Ambulatory stroke patients; Gait training; Lokomat; Physical therapy
MeSH Terms: conditions — Stroke; Infarction, Middle Cerebral Artery

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- A-B (Experimental): Gait training by an automatic gait trainer (Lokomat) for 3 weeks followed by 3 weeks of categorized gait training by a physical therapist
  Interventions: Behavioral: Lokomat - Physical therapy
- B-A (Experimental): Categorized gait training by physical therapists for 3 weeks followed by 3 weeks of lokomat training
  Interventions: Behavioral: Physical therapy - Lokomat

INTERVENTIONS:
Behavioral: Lokomat - Physical therapy — A: Lokomat training, 30 minutes per day for 3 weeks, 5 days per week. B: Categorized gait training by physical therapist, 30 minutes per day for 3 weeks, 5 days per week
  Arms: A-B
Behavioral: Physical therapy - Lokomat — B: Daily 30 minutes of gait training with a physical therapist, 5 days per week for 3 weeks.
  A: Daily 30 minutes of Lokomat training, 5 days per week for 3 weeks.
  Arms: B-A

SUMMARY:
The objective of this study is to investigate the effects of an automatic gait trainer (Lokomat) handled by physical therapists compared with categorized gait training by physical therapists in ambulatory stroke patients. Gait speed, gait distance and gait symmetry are used to evaluate study effects.

Hypotheses: 1) The Lokomat improves stroke patients gait speed, distance and symmetry more than categorized gait training.

ELIGIBILITY:
Inclusion Criteria:

1. First time Stroke
2. Middle cerebral artery infarction
3. Less than three month from stroke onset
4. Able to walk with or without a stick at gait speed less than 0.5 m/s
5. Participants are able to cope with the Lokomat

Exclusion Criteria:

1. Co-morbidity which impedes study participations
2. Language deficits which makes it impossible to understand oral or written study instructions
3. More than 190 cm tall and 135 kg in weight
4. Pregnancy
5. No gait function prior stroke
6. Skin sore or eruption on lower extremity or trunk, differences in lower extremity length of more than 2 cm or contracture of lower extremity which impedes gait training in the Lokomat -

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2007-06; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
10 meters walking test (gait speed) | at inclusion, week 3 and week 6

SECONDARY OUTCOMES:
Six minutes walking test | Inclusion, wek 3 and week 6
Gait symmetry index | Inclusion, week 3 and week 6
Timed Up And Go | Inclusion, Week 3 and Week 6

CONTACTS AND LOCATIONS:
Overall Officials: Jørgen F Nielsen, Professor, Study Chair — Hammel Neurorehabilitation and Research Center, Denmark; Carsten Kock-Jensen, MD, Study Director — Hammel Neurorehabilitation and Research Center, Denmark; John Brincks, PhD student, Principal Investigator — Hammel Neurorehabilitation and Reseach Center
Locations (1):
- Hammel Neurorehabilitation and Research Center, Hammel, Denmark